CLINICAL TRIAL: NCT00514696
Title: Open Label Phase 2 Study of the Safety and Biological Activity of GCS-100 in Subjects With Chronic Lymphocytic Leukemia
Brief Title: Study of the Safety of GCS-100 in Subjects With Chronic Lymphocytic Leukemia
Acronym: PR-CS008
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-CS008
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Cancer; Leukemia; GCS-100; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms; Leukemia | interventions — GCS-100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GCS-100 (Experimental): GCS-100: 160 mg/m2 IV (in the vein) Study Days 1-5 of each 21-day cycle
  Interventions: Drug: GCS-100

INTERVENTIONS:
Drug: GCS-100 — GCS-100: 160 mg/m2 IV (in the vein) Study Days 1-5 of each 21-day cycle

SUMMARY:
The purpose of this study is to evaluate the safety of GCS-100 and the biologic activity of GCS-100 in subjects with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety of GCS-100, and effect of GCS-100 on markers of apoptosis in subjects with chronic lymphocytic leukemia. The secondary objective of this study is to evaluate the effect of GCS-100 on peripheral blood leukocyte count in subjects with chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must meet all of the following criteria:

1. Subject is capable of understanding the purpose and risks of the study and is able to provide written Informed Consent.
2. Subject is male or female, aged at least 18 years.
3. Subject has been diagnosed with chronic lymphocytic leukemia.
4. Subject has Stage II or higher, chronic lymphocytic leukemia that currently requires therapy due to the severity of the disease symptoms and/or to the presence of increasing anemia and/or increasing splenomegaly.
5. Subject has received 2 or fewer prior therapies for his/her chronic lymphocytic leukemia.
6. Subject does not currently require blood transfusions.
7. Subject's peripheral blood leukocyte count is > 10,000 cells/mm3.
8. Subject's Karnofsky performance status is > 60%.
9. Subject's life expectancy is at least 3 months.
10. Female subjects of childbearing potential (i.e., women who have not been surgically sterilized or have not been post-menopausal for at least 1 year), and male subjects with partners of childbearing potential, must agree to use medically acceptable methods of contraception throughout the entire study period.
11. Subject is willing and able to comply with the prescribed treatment protocol and evaluations.

Exclusion Criteria:

Subjects will be ineligible for study participation if they meet any of the following criteria:

1. Subject received biologic therapy and/or chemotherapy that may be active against chronic lymphocytic leukemia within the 4 weeks prior to Study Day 1.
2. Subject is anticipated to require steroid therapy within the next 21 days.
3. Subject received an investigational (i.e., experimental) therapy within the 4 weeks prior to Study Day 1.
4. Subject's clinical laboratory values meet any of the following criteria within the 7 days prior to Study Day 1:

   * Platelet count < 25,000 cells/mm3
   * Absolute neutrophil count < 500 cells/mm3
   * Hemoglobin < 8.0 g/dL and with an autoimmune hemolytic component to the subject's anemia
   * AST and/or ALT > 2.5 X the upper limit of normal
   * Total bilirubin > 1.5 X the upper limit of normal
   * Serum creatinine > 2 mg/dL
5. Subject has a known history of human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C infection.
6. Subject has a clinically relevant active infection and/or a serious co-morbid medical condition, such as recent myocardial infarction, unstable angina, difficult-to-control congestive heart failure, uncontrolled hypertension, difficult-to-control cardiac arrhythmias, chronic obstructive or chronic restrictive pulmonary disease, cirrhosis, inflammatory bowel disease.
7. Subject had major surgery within the 4 weeks prior to Study Day 1.
8. Subject had another malignancy within the 3 years prior to study entry, with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer, or other cancer for which the subject has been disease-free for at least 3 years.
9. If female, subject is pregnant or breast-feeding.
10. Subject has a concomitant disease or condition, including laboratory abnormalities, which in the opinion of the Investigator could interfere with the conduct of the study or could put the subject at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To Evaluate the effect of GCS-100 on markers of apoptosis in subjects with chronic lymphocytic leukemia using physical examinations, vital signs, lab assessments, and adverse event reporting | Up to 15 cycles X 21 days

SECONDARY OUTCOMES:
To evaluate the effect of GCS-100 on peripheral blood leukocyte count in subjects with chronic lymphocytic leukemia using complete blood count, leukocyte count and circulating cells for apoptosis | Hour 6 after Day 1 dosing, and Days 4 and 8

CONTACTS AND LOCATIONS:
Overall Officials: David Smith, MD, Principal Investigator — US Oncology
Locations (8):
- United States (8):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Cancer Centers of Florida, Winter Park, Florida
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Dayton Oncology & Hematology, Kettering, Ohio
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists - Vancouver Cancer Center, Vancouver, Washington
  - Yakima Cancer Center, Yakima, Washington